CLINICAL TRIAL: NCT02440165
Title: Basic Care Revisited: an Early Nursing Nutrition Intervention for Outpatients in Need of Surgery
Brief Title: Basic Care Revisited: Early Nutrition Intervention for Outpatients
Acronym: BCR_N
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014-1353
Record Dates: First submitted 2015-03-11; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Malnutrition; Dietary Modification
Keywords: nutrition; nurse; intervention; malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): The early nursing nutrition intervention will include malnutrition screening (during outpatient clinic visit) with the MUST. If patients are ´at risk for malnutrition´ or ´malnourished´, a standardized nutrition care plan will be discussed with the patient by the nurse. This nutrition care plan will include:
  * Information and advice;
  * Examples of energy and protein rich meals;
  * patients will be asked to register their nutritional intake for two days at home;
  * after a week, the nurse will call the patients to answer questions and to give advice.
  This nutrition care plan will be tailored to the individual patient requirements.
  Furthermore, if patients are 'malnourished', a visit to the dietician is always suggested, because this is usual care.
  Interventions: Behavioral: Nursing nutrition intervention
- Usual care (No Intervention): All participants, both in the intervention group and the control group, receive usual care containing a regular visit to a nurse who will perform a malnutrition screening with the MUST (Malnutrition Universal Screening Tool). If patients are 'malnourished', a visit to the dietician is suggested.

INTERVENTIONS:
Behavioral: Nursing nutrition intervention — The early nursing nutrition intervention will include malnutrition screening (during outpatient clinic visit) with the MUST. If patients are ´at risk for malnutrition´ or ´malnourished´, a standardized nutrition care plan will be discussed with the patient by the nurse. This nutrition care plan will include:
  * Information and advice;
  * Examples of energy and protein rich meals;
  * patients will be asked to register their nutritional intake for two days at home;
  * after a week, the nurse will call the patients to answer questions and to give advice.
  This nutrition care plan will be tailored to the individual patient requirements.
  Furthermore, if patients are 'malnourished', a visit to the dietician is always suggested, because this is usual care.
  Arms: Experimental

SUMMARY:
Early nursing nutrition intervention for outpatients in need of surgery

* Objective - To investigate the feasibility and effectiveness of screening and an early nursing intervention on malnutrition in outpatients in need for surgery.
* Design - Multi-centre cluster-randomised controlled early trial design (n=150 patients)
* Intervention - Malnutrition screening (during outpatient clinic visit) and (in case of patients being ´at risk for malnutrition´ or being ´malnourished´), a nutrition care plan (including nutritional drinks and energy and protein rich meals) tailored to individual patient requirements
* Comparison - Usual care (no nutritional care plan)

DETAILED DESCRIPTION:
Early screening and treatment of malnutrition is vital. The prevalence of malnutrition at hospital admission has only slightly decreased over the last few years. (Halfens, 2007) This indicates that screening and intervention early in the course of developing disease, e.g. at the outpatient clinic, can prevent severe malnutrition and decrease the amount and complexity of care. (Jonkers-Schuitema et al., 2011; Leistra et al., 2009). Screening for malnutrition and nutrition interventions at the outpatient clinic however, is no daily practice. Leistra et al. (2009) showed that only 17% of the severely undernourished patients and 4% of the moderately undernourished patients received some form of dietetic treatment at the outpatient clinic. Early nursing nutrition interventions have not been studies well before.

Aim: To investigate the feasibility and effectiveness of screening and an early nursing intervention on malnutrition in outpatients in need for surgery.

Design: Multicentre cluster randomized controlled trial design in surgical outpatient clinics in two hospitals (one academic and one non-academic). The intervention is randomly assigned to half of the outpatient clinics, and patients clustered with these nurses, working at the outpatient clinics. The remaining nurses and their patients will serve as a control group. Nursing teams with nurses working in multiple teams will be excluded. Nurses will be trained in the use of the MUST-Screening and nutrition care plans. Study population: Patients visiting the outpatient clinic, planned for operation, of one academic and one non-academic hospital (n=150).

Description of the intervention: The early nursing nutrition intervention will include malnutrition screening (during outpatient clinic visit) with the MUST. If patients in the intervention group are being ´at risk for malnutrition´ or being ´malnourished´, a standardised nutrition care plan (including nutritional drinks and energy and protein rich meals, tailored to individual patient requirements) will be discussed with the patient by nurses. Control patients will receive usual care (no nutrition care plan). The intervention period will be 6 months.

Outcome: Primary: Up to 6 months, BMI will be measured at three point in time: 1) at the outpatient clinic, 2) at hospitalisation, and 3) at discharge. Also, intake of nutrients will be measured for 2 days after the outpatient clinic visit. Average time frame for each patient is 5 weeks, for both intervention and control group.

Secondary: Up to 6 months, Length of Stay (LOS) and health-related quality of life (EQ-5D) will be measured at discharge, and CQ satisfaction with nutritional care & care in general will be measured at the outpatient clinic and at hospitalisation. Average time frame for each patient is 5 weeks, for both intervention and control group.

To evaluate costs of the intervention, nurses time investment with patients at risk will be observed in 30 patients per group and combined with average costs to arrive at a preliminary cost of usual care and the early nutrition intervention. To evaluate the process, nurses will be interviewed (n=6) to collect data on the manner in which the intervention changes the nursing care.

Statistical analysis: Data will be analysed on an intention-to-treat basis. Results are clustered at ward level. In this study with the same subjects at baseline and follow-up, we will therefore use a linear mixed model for repeated measurements, with ''nurse'' as random effect, BMI as main outcome, and group, time and the group x time interaction as fixed effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for surgery within 6 weeks after the outpatient clinic visit;
* Patients with an age of 18 years or older;
* Patients with the ability to speak and read the Dutch language.

Exclusion Criteria:

* Hospital admission within one week after the outpatient clinic visit;
* Expected hospital admission < 5 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in BMI | Up to 6 months
  body mass index: at 3 points in time; 1) at the outpatient clinic, 2) at hospitalisation, and 3) at discharge. Average time frame for each patient is 5 weeks.

SECONDARY OUTCOMES:
LOS | Up to 6 months
  Length of hospital stay: at discharge
Health related QoL | Up to 6 months
  Health related Quality of life: at discharge
CQ satisfaction | Up to 6 months
  after outpatient clinic visit, and at hospitalisation: Satisfaction in general for 'Nursing care' and specified for nutritional care. This question is derived from the Consumer Quality Index (http://www.centrumklantervaringzorg.nl/publicaties/publicaties-cq-index.html)
Costs | Up to 6 months
  To evaluate costs of the intervention, the reach and delivery data collected for the purpose of process evaluation will be used, and combined with cost estimates for both the intervention and usual care, from the perspective of direct healthcare costs. In the analysis the outcomes of the intervention and care as usual (specific and generic outcomes) will be matched with the costs of implementation, costs of nursing care performed (in euros per hour, observed in 30 patients per group) and costs of training and materials. In this way a first exploration of cost effectiveness will be available.
Process | Up to 6 months
  An adapted version of the Linnan and Steckler framework for conducting process evaluation studies will be used (Linnan and Steckler, 2002, Saunders et al., 2005).

CONTACTS AND LOCATIONS:
Overall Officials: Ria Nijhuis- van der Sanden, PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Sint Maartenskliniek, Nijmegen, Gelderland
  - Radboudumc, Nijmegen, Gelderland

REFERENCES:
- [Derived] van Noort HHJ, Witteman BJM, Vermeulen H, Huisman-de Waal G; Basic Care Revisited research group. An outpatient nursing nutritional intervention to prehabilitate undernourished patients planned for surgery: A multicentre, cluster-randomised pilot study. Clin Nutr. 2020 Aug;39(8):2420-2427. doi: 10.1016/j.clnu.2019.11.038. Epub 2019 Dec 2. PMID 31879076